CLINICAL TRIAL: NCT06533345
Title: MERCI Chronic Pain Research Clinic (Medical Education and Research in Compassionate Integration/Intervention)
Brief Title: VCOM Pain Free Research
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Edward Via Virginia College of Osteopathic Medicine (Other)
Responsible Party: Principal Investigator, William Pearson, Discipline Chair for Anatomy, Edward Via Virginia College of Osteopathic Medicine
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2024--061
Record Dates: First submitted 2024-07-19; First posted 2024-08-01 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Chronic Pain
Keywords: Autonomic Dysfunction; Sympathetic Dominance; Osteopathic Manipulative Treatment; Dry Needling; Nutrition; Lifestyle; Group Therapy; Therapy; Trauma; Flourishing
MeSH Terms: conditions — Chronic Pain; Primary Dysautonomias; Wounds and Injuries | interventions — Nutritional Status; Dry Needling; Manipulation, Osteopathic

STUDY DESIGN:
Intervention Model Description: This research is a prospective longitudinal observational study to gather preliminary data for a future Sequential Multiple Assignment Randomized Trial (SMART).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Osteopathic Manipulative Treatment (Experimental): Osteopathic Manipulative Treatment
  Interventions: Other: Osteopathic Manipulative Treatment
- Dry Needling (Experimental): Dry Needling
  Interventions: Procedure: Dry Needling
- Autonomic Recalibration (Experimental): Autonomic Recalibration
  Interventions: Other: Autonomic Recalibration
- Nutrition (Experimental): Nutrition
  Interventions: Behavioral: Nutrition
- Behavior Change Coaching (Experimental): Behavior Change Coaching
  Interventions: Behavioral: Behavior Change Coaching
- Counseling Psychology (Experimental): Counseling Psychology
  Interventions: Behavioral: Counseling Psychology
- Multiple (Experimental): Multiple
  Interventions: Behavioral: Behavior Change Coaching; Behavioral: Nutrition; Other: Autonomic Recalibration; Procedure: Dry Needling; Other: Osteopathic Manipulative Treatment; Behavioral: Counseling Psychology; Other: Multiple Treatments

INTERVENTIONS:
Behavioral: Behavior Change Coaching — Done by Dr. Hollingsworth or students via consultations with participants. Participant's health behavior aspirations or target outcomes will be clarified, informed by the participant's interactions with other MERCI providers. Behaviors that move the participant towards their aspirations/outcomes will be explored to find target behaviors that the participant is motivated and able to do. Target behaviors and supporting habits will be designed into the participant's existing routine. The Fogg Behavior Model will be used 1) to find the participant's primary motivation for engaging in target behaviors and 2) to make target behaviors easier to do. Implementation intentions - When/then or If/then plans - will be used to form habits and promote behavior engagement. Adopting a growth mindset will also be discussed. Subsequent consultations will focus on troubleshooting, iterative improvements, and incorporation of new aspirations/outcomes, target behaviors, and supporting habits.
  Arms: Behavior Change Coaching; Multiple
Behavioral: Nutrition — Nutrition: The nutrition intervention will be conducted as a 12-week protocol with assessment points at baseline, 1 month, and 3 months. Following consent, eligible participants will work through a self-taught educational module detailing the anti-inflammatory dietary program. Once the module is completed, participants will be scheduled for one-on-one counseling sessions with a Registered Dietitian or a supervised Dietetic Intern or Medical Student on the research team to receive personalized guidance on implementation of the dietary intervention. A dietary recall will be conducted via the automated self-administered dietary assessment tool (ASA24®), which takes about 20 minutes to complete. This survey will be conducted on two non-consecutive days at each timepoint (baseline, 1 month, and 3 months).
  Arms: Multiple; Nutrition
Other: Autonomic Recalibration — Participant will be outfitted with the Empatica wrist sensor. An initial history to rule out pathology and document a chief complaint relevant to pain is conducted. An initial head to toe assessment of withdrawal or startle reflex behavior in response to palpation is performed to identify trigger points and establish patterns of sympathetic dominance. The pattern of sympathetic dominance is addressed during treatment by Primal Reflex Release Technique Protocol to inhibit somatic afferent feedback loops and rebalance the autonomic nervous system towards a state of parasympathetic dominance. Day 2 is the same until the initial history and r/o. Here, the history is from the previous day, asking about perception of pain, sleep, digestion, or other pertinent issues brought up on the first visit. Treatment proceeds same as Day 1. Any emotional tags to trigger points are identified and acknowledged. Subjects may be scheduled for follow-up visits if their pain persists.
  Arms: Autonomic Recalibration; Multiple
Procedure: Dry Needling — An initial history to document a chief complaint relevant to pain is conducted and to identify and potential contraindications (infection of overlying skin, patient on anticoagulation drugs, 1st trimester of pregnancy, etc.) A physical exam is performed to identify the trigger points causing pain. The subject is educated about the risks/benefits/indications and alternative treatments. The subject is also educated about dry needling aftercare. The skin over the trigger points is cleaned with 70% isopropyl alcohol. The pertinent trigger points are treated with dry needling (95% of time), direct inhibition (2 - 3% of time) or injection of 1% lidocaine in a fan-like fashion (1 - 2 % of the time). Subject is assessed for any bleeding. An office note, including a procedure note, is documented in the subject's record. Subject is scheduled for additional follow-up meeting.
  Arms: Dry Needling; Multiple
Other: Osteopathic Manipulative Treatment — Osteopathic Manipulative Treatment: After inform and consent process, the subject will enter patient room and meet with Dr. Hayes, who will conduct a brief history of patient pain, injuries, and procedures. Subjects will be asked to wear, or change into, athletic shorts or a tank top or loose-fitting T-shirt to facilitate treatment. Subject will undergo a brief somatic dysfunction screen, which involves light tough and manipulation. Once Hayes has diagnosed potential dysfunctions, he will proceed with osteopathic manipulative treatment. Treatment will last anywhere from 15 minutes to 1 hour. At the end of the treatment, subjects will be scheduled for a follow-up visit.
  Arms: Multiple; Osteopathic Manipulative Treatment
Behavioral: Counseling Psychology — Psychoeducation Workshop and Counseling: The psychoeducational group intervention will be done according to the standardized Empowered Relief (Darnall et al., 2024) protocol. Empowered Relief is a single-session, 2-hour group workshop (online or in person) that teaches participants pain neuroscience education, mindfulness principles, and cognitive-behavioral skills. During the program, participants will complete a personalized plan to work toward pain relief. This program requires a certified instructor; Marilyn Cornish (Co-I), a licensed psychologist, is certified. After completion, participants can attend up to 4 individual counseling sessions with a counseling psychology doctoral student (supervised by Marilyn Cornish). Sessions will be approximately 50-60 minutes and will occur every other week. Specific in-session interventions will be tailored to the participant's unique needs but will focus on participants' pain relief plan and overall psychological wellbeing of participants.
  Arms: Counseling Psychology; Multiple
Other: Multiple Treatments — Subjects receiving multiple treatment interventions over the same period of time.
  Example: A subject joins the Osteopathic Manipulative Treatment group and meets with Dr. Hayes for treatment visits. At the same time, they are meeting with Dr. Kirby in a separate visit (or at the same time, if scheduling allows) to discuss Nutrition. Any subjects who were in multiple/overlapping treatment groups will fit this description.
  Arms: Multiple

SUMMARY:
Studies estimate that 30% of people worldwide experience chronic pain. The mechanisms causing this pain can vary: a neuropathic offender, such as nerve compression; a structural offender, such as long-term effects of soft tissue damage and repair; or nociplastic, dysfunctional offenders, such as fibromyalgia. The type of pain experienced influences diagnostic and treatment choice. In theory, there's a significant blending of these pain types within individuals and across patients, leading many specialists to view pain classification as a spectrum. Multidisciplinary pain management (MPM) is a standard model for addressing and treating different mechanisms of chronic pain using multiple interventions from different disciplines. Although many clinics employing these strategies have resulted in positive and clinically effective outcomes, the creation and implementation of such facilities have not been widespread. With increasing focus on psychosocial factors that impact pain in conjunction with structural and biomechanical offenders, a need for a whole-person, integrated approach to chronic pain management is needed. We propose an observational study to gather data that will inform the design, implementation, and operation of such a chronic pain research clinic.

ELIGIBILITY:
Inclusion Criteria:

* Those experiencing chronic pain, i.e., ongoing pain not relevant to an acute perturbation (e.g., recent injury).

Exclusion Criteria:

* Those subjects seeking pharmaceutical intervention
* Those whose myofascial pain is deemed functional (normal response to acute injury or ongoing pathology

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-08-30 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity (NRS Pain Scale) | Beginning of each Visit through study completion, an average (anticipated) of 6 months
  0-10 Pain Rating. 0=no pain to 10=pain as intense as you can imagine
PROMIS (Pain Interference, SF4a) | Beginning of each Visit through study completion, an average (anticipated) of 6 months
  Pain interference survey. Answers range from "Not at all" to "Very Much" when relating to the impact of pain on daily life.
Use of analgesics (QAQ-Quantitative Analgesic Questionnaire) | Beginning of each Visit through study completion, an average (anticipated) of 6 months
  Survey listing all medications taken for pain. All types are converted in equivalent doses of morphine and scored.
Human Flourishing (Secure Flourishing Index) | Beginning of each Visit through study completion, an average (anticipated) of 6 months
  Measure of Human Flourishing across 6 Domains. Scores range from 0-10 with lower scores indicating lower flourishing and higher scores indicating higher flourishing.

CONTACTS AND LOCATIONS:
Locations (1):
- Edward Via College of Osteopathic Medicine-Auburn, Auburn, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kuntz JL, Young DR, Saelens BE, Frank LD, Meenan RT, Dickerson JF, Keast EM, Fortmann SP. Validity of the Exercise Vital Sign Tool to Assess Physical Activity. Am J Prev Med. 2021 Jun;60(6):866-872. doi: 10.1016/j.amepre.2021.01.012. Epub 2021 Mar 27. PMID 33781618
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Barkham, Michael, Bewick, Bridgette, Mullin, Tracy, Gilbody, Simon, Connell, Janice, Cahill, Jane, Mellor-Clark, John, Richards, David, Unsworth, Gisela, Evans, Chris, (2013), The CORE-10: A short measure of psychological distress for routine use in the psychological therapies. Counselling and Psychotherapy Research, 13 doi: 10.1080/14733145.2012.729069.
- [Background] Sullivan, M. J. L., Bishop, S. R., & Pivik, J. (1995). The Pain Catastrophizing Scale: Development and validation. Psychological Assessment, 7(4), 524-532. https://doi.org/10.1037/1040-3590.7.4.524
- [Background] Hooper, L. M., Stockton, P., Krupnick, J., & Green, B. L. (2011). The development, use, and psychometric properties of the Trauma History Questionnaire. Journal of Loss and Trauma, 16, 258-283.
- [Background] Jensen, Mark P., Hypnosis for Chronic Pain Management: Therapist Guide, Treatments That Work (New York, 2011; online edn, Oxford Academic, 1 Apr. 2015), https://doi.org/10.1093/med:psych/9780199772377.001.0001, accessed 12 Mar. 2024.
- [Background] Robinson-Papp J, George MC, Wongmek A, Nmashie A, Merlin JS, Ali Y, Epstein L, Green M, Serban S, Sheth P, Simpson DM. The Quantitative Analgesic Questionnaire: A Tool to Capture Patient-Reported Chronic Pain Medication Use. J Pain Symptom Manage. 2015 Sep;50(3):381-6. doi: 10.1016/j.jpainsymman.2015.03.013. Epub 2015 Apr 23. PMID 25912277
- [Background] Amtmann D, Cook KF, Jensen MP, Chen WH, Choi S, Revicki D, Cella D, Rothrock N, Keefe F, Callahan L, Lai JS. Development of a PROMIS item bank to measure pain interference. Pain. 2010 Jul;150(1):173-182. doi: 10.1016/j.pain.2010.04.025. PMID 20554116
- [Background] Felitti VJ, Anda RF, Nordenberg D, Williamson DF, Spitz AM, Edwards V, Koss MP, Marks JS. Relationship of childhood abuse and household dysfunction to many of the leading causes of death in adults. The Adverse Childhood Experiences (ACE) Study. Am J Prev Med. 1998 May;14(4):245-58. doi: 10.1016/s0749-3797(98)00017-8. PMID 9635069
- [Background] Edwards LC, Pearce SA, Turner-Stokes L, Jones A. The Pain Beliefs Questionnaire: an investigation of beliefs in the causes and consequences of pain. Pain. 1992 Dec;51(3):267-272. doi: 10.1016/0304-3959(92)90209-T. PMID 1491853
- [Background] Vartiainen P, Heiskanen T, Sintonen H, Roine RP, Kalso E. Health-related quality of life change in patients treated at a multidisciplinary pain clinic. Eur J Pain. 2019 Aug;23(7):1318-1328. doi: 10.1002/ejp.1398. Epub 2019 May 3. PMID 30980782
- [Background] Kress HG, Aldington D, Alon E, Coaccioli S, Collett B, Coluzzi F, Huygen F, Jaksch W, Kalso E, Kocot-Kepska M, Mangas AC, Ferri CM, Mavrocordatos P, Morlion B, Muller-Schwefe G, Nicolaou A, Hernandez CP, Sichere P. A holistic approach to chronic pain management that involves all stakeholders: change is needed. Curr Med Res Opin. 2015;31(9):1743-54. doi: 10.1185/03007995.2015.1072088. Epub 2015 Aug 20. PMID 26172982
- [Background] Asmundson GJ, Katz J. Understanding the co-occurrence of anxiety disorders and chronic pain: state-of-the-art. Depress Anxiety. 2009;26(10):888-901. doi: 10.1002/da.20600. PMID 19691031
- [Background] Cohen SP, Vase L, Hooten WM. Chronic pain: an update on burden, best practices, and new advances. Lancet. 2021 May 29;397(10289):2082-2097. doi: 10.1016/S0140-6736(21)00393-7. PMID 34062143
- [Background] Seton B, Pandey R, Piscura MK, Pearson WG Jr. Autonomic Recalibration: A Promising Approach for Alleviating Myofascial Pain Explored in a Retrospective Case Series. Cureus. 2024 Jan 17;16(1):e52450. doi: 10.7759/cureus.52450. eCollection 2024 Jan. PMID 38371140
- [Background] Charles D, Hudgins T, MacNaughton J, Newman E, Tan J, Wigger M. A systematic review of manual therapy techniques, dry cupping and dry needling in the reduction of myofascial pain and myofascial trigger points. J Bodyw Mov Ther. 2019 Jul;23(3):539-546. doi: 10.1016/j.jbmt.2019.04.001. Epub 2019 Apr 4. PMID 31563367
- [Background] Clar C, Tsertsvadze A, Court R, Hundt GL, Clarke A, Sutcliffe P. Clinical effectiveness of manual therapy for the management of musculoskeletal and non-musculoskeletal conditions: systematic review and update of UK evidence report. Chiropr Man Therap. 2014 Mar 28;22(1):12. doi: 10.1186/2045-709X-22-12. PMID 24679336
- [Background] Mejia-Mejia E, Budidha K, Abay TY, May JM, Kyriacou PA. Heart Rate Variability (HRV) and Pulse Rate Variability (PRV) for the Assessment of Autonomic Responses. Front Physiol. 2020 Jul 23;11:779. doi: 10.3389/fphys.2020.00779. eCollection 2020. PMID 32792970
- [Background] Darnall BD, Burns JW, Hong J, Roy A, Slater K, Poupore-King H, Ziadni MS, You DS, Jung C, Cook KF, Lorig K, Tian L, Mackey SC. Empowered Relief, cognitive behavioral therapy, and health education for people with chronic pain: a comparison of outcomes at 6-month Follow-up for a randomized controlled trial. Pain Rep. 2024 Jan 25;9(1):e1116. doi: 10.1097/PR9.0000000000001116. eCollection 2024 Jan. PMID 38288134
- [Background] Evans C, Connell J, Barkham M, Margison F, McGrath G, Mellor-Clark J, Audin K. Towards a standardised brief outcome measure: psychometric properties and utility of the CORE-OM. Br J Psychiatry. 2002 Jan;180:51-60. doi: 10.1192/bjp.180.1.51. PMID 11772852
- [Background] Sullivan MJL, Bishop SR and Pivik J. The Pain Catastrophizing Scale: development and validation. Psychological assessment. 1995;7(4):524-532